CLINICAL TRIAL: NCT05054036
Title: Efficacy, Safety, and Tolerability of MoviPrep® Versus GoLYTELY® Bowel Preparation in Hospitalized Patients Undergoing Colonoscopy: a Randomized Control Trial
Brief Title: MoviPrep® Versus GoLYTELY® Bowel Preparation in Hospitalized Patients Undergoing Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000031169; 000 (Other: CTGTY)
Record Dates: First submitted 2021-09-09; First posted 2021-09-23 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Bowel Preparation Before Colonoscopy
Keywords: colonoscopy; bowel preparation; inpatient; tolerability
MeSH Terms: interventions — MoviPrep; Golytely

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MoviPrep (Experimental): For MoviPrep, the dose, schedule, and route of administration are as follows:
  * On the evening prior to the colonoscopy, mix the powder with lukewarm water to a total volume of 32 oz. Drink 8 oz. every 15 minutes until the solution is finished. Drink 16 oz. of clear liquids before bed.
  * On the morning of the procedure, repeat the above steps and make sure all fluids are consumed at least 2 hours prior to colonoscopy.
  * Limit food intake to a regular breakfast, light lunch and clear soup or plain yogurt for dinner on the day prior to the colonoscopy (completed at least 1 hour prior to the first MoviPrep dose.
  * Consume only clear liquids from the start of MoviPrep until after the colonoscopy.
  Interventions: Drug: MoviPrep
- GoLYTELY (Active Comparator): For GoLYTELY, the dose, schedule, and route of administrate are as follows:
  * On the evening prior to the colonoscopy, mix powder with lukewarm water to a total volume of 4 liters. Drink 2 liters of the solution and store the rest in the refrigerator.
  * Drink the remaining 2 liters on the morning of the procedure.
  * Limit food intake to a light breakfast on the day prior to the colonoscopy, followed by only clear liquids until the procedure is complete.
  * Avoid red and purple liquids.
  Interventions: Drug: Golytely

INTERVENTIONS:
Drug: MoviPrep — Split-dose MoviPrep bowel preparation
  Arms: MoviPrep
Drug: Golytely — Split-dose GoLYTELY bowel preparation
  Arms: GoLYTELY

SUMMARY:
Adequate bowel cleansing is a critical component in the care of hospitalized patients undergoing colonoscopy. However, inpatient status is a well-established risk factor for inadequate bowel preparation. However, few strategies have been rigorously shown to reduce the risk of inadequate bowel preparation. Moreover, inadequate bowel preparation is frequently related to the poor tolerability of high volumes of bowel preparation in the medically complex and comorbid hospitalized population. Low volume bowel preparations have been developed that have been shown to be noninferior compared to high volume bowel preparation with regards to adequacy of bowel preparation but with improved tolerability. However, the use of low volume bowel preparations for colonoscopies have largely been evaluated in the outpatient setting. In this study, we plan to compare rates of adequate bowel preparation and tolerability of a low volume bowel preparation, MoviPrep, compared to standard high volume bowel preparation, GoLYTELY, in hospitalized patients undergoing colonoscopy. This study promises to highlight low volume bowel preparation as a viable and better tolerated alternative to high volume bowel preparation in hospitalized patients which may ultimately decrease delays in inpatient endoscopy as well as hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or greater
4. Hospitalized patient scheduled to undergo colonoscopy with bowel preparation (not including preparation with enemas alone)
5. Ability to take bowel preparation and be willing to adhere to the regimen

Exclusion Criteria:

1. Patients presenting to the hospital with ileus, toxic megacolon, evidence of gastrointestinal obstruction
2. Receipt of bowel preparation for other reasons during their hospitalization prior to their colonoscopy
3. Patients with prior significant gastrointestinal surgeries including colonic resection, subtotal colectomy, abdomino-perineal resection, Hartmann's procedure or other similar surgeries involving structure/function of small intestine or colon
4. Unable to give informed consent to the procedure
5. Known glucose-6-phosphate dehydrogenase deficiency
6. Known phenylketonuria
7. Known hypersensitivity to polyethylene glycols or ascorbic acid
8. Patients undergoing colonoscopy for foreign body removal and/or decompression
9. Pregnancy or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Score (BBPS) During Colonoscopy Withdrawal | At time of procedure, approximately 45 minutes
  The BBPS is a validated scoring tool that assesses the three segments of the colon (left, transverse, right) and rates them from 1-3 based on the ability to visualize the mucosa. An adequate bowel preparation is defined as a BBPS of 6 or higher with no individual segment scoring less than a 2.

SECONDARY OUTCOMES:
Mayo Clinic Bowel Preparation Questionnaire | Immediately prior to procedure
  The Mayo Clinic Bowel Preparation Questionnaire is a survey consisting of 9 questions that relate to symptoms and tolerability of bowel preparation before colonoscopy. The answers to each question will be aggregated for each arm and compared.
BBPS Score During Colonoscopy Withdrawal For Each Segment | At time of procedure, approximately 45 minutes
  BBPS assesses three segments of the colon (left, transverse, right) and rates each segment either a 1, 2, or 3 based on the ability to visualize the mucosa. Higher scores correspond to improved mucosal visibility.
Rates of "Excellent" Bowel Preparation | At time of procedure, approximately 45 minutes
  The BBPS is a validated scoring tool that assesses the three segments of the colon (left, transverse, right) and rates them from 1-3 based on the ability to visualize the mucosa. An excellent bowel preparation is defined as a BBPS score of an 8 or 9.
Cecal Intubation Rate | At time of procedure, approximately 45 minutes
  Percentage of colonoscopies during which the cecum is successfully reached
Cecal Intubation Time | At time of procedure, approximately 45 minutes
  Time from insertion of colonoscopy to reaching the cecum
Colonoscopy Withdrawal Time | At time of procedure, approximately 45 minutes
  Time from reaching the cecum to complete withdrawal of the colonoscope
Time to Endoscopy | At time of procedure, approximately 45 minutes
  The time from when the patient started the bowel preparation to the colonoscopy procedure itself.
Hospital Length of Stay | After study completion, an average of 5 days
  Time from admission to discharge
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Through study completion, an average of 3 days
  The National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term from a scale of 1-5, with increasing score corresponding to increasing AE severity.

CONTACTS AND LOCATIONS:
Overall Officials: Darrick K Li, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale New-Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadlapati R, Johnston ER, Gregory DL, Ciolino JD, Cooper A, Keswani RN. Predictors of Inadequate Inpatient Colonoscopy Preparation and Its Association with Hospital Length of Stay and Costs. Dig Dis Sci. 2015 Nov;60(11):3482-90. doi: 10.1007/s10620-015-3761-2. Epub 2015 Jun 21. PMID 26093612
- [Background] Fuccio L, Frazzoni L, Spada C, Mussetto A, Fabbri C, Manno M, Aragona G, Zagari RM, Rondonotti E, Manes G, Occhipinti P, Cadoni S, Bazzoli F, Hassan C, Radaelli F; QIPS study group. Factors That Affect Adequacy of Colon Cleansing for Colonoscopy in Hospitalized Patients. Clin Gastroenterol Hepatol. 2021 Feb;19(2):339-348.e7. doi: 10.1016/j.cgh.2020.02.055. Epub 2020 Mar 18. PMID 32200083
- [Background] Spadaccini M, Frazzoni L, Vanella G, East J, Radaelli F, Spada C, Fuccio L, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Van Hooft JE, Dumonceau JM, Marmo C, Alfieri S, Chandrasekar VT, Sharma P, Rex DK, Repici A, Hassan C. Efficacy and Tolerability of High- vs Low-Volume Split-Dose Bowel Cleansing Regimens for Colonoscopy: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2020 Jun;18(7):1454-1465.e14. doi: 10.1016/j.cgh.2019.10.044. Epub 2019 Nov 1. PMID 31683057
- [Background] Garber A, Sarvepalli S, Burke CA, Bhatt A, Ibrahim M, McMichael J, Morris-Stiff G, Rizk MK, Vargo JJ, Rothberg MB. Modifiable Factors Associated with Quality of Bowel Preparation Among Hospitalized Patients Undergoing Colonoscopy. J Hosp Med. 2019 May;14(5):278-283. doi: 10.12788/jhm.3173. PMID 30986186
- [Background] Patel M, Staggs E, Thomas CS, Lukens F, Wallace M, Almansa C. Development and validation of the Mayo Clinic Bowel Prep Tolerability Questionnaire. Dig Liver Dis. 2014 Sep;46(9):808-12. doi: 10.1016/j.dld.2014.05.020. Epub 2014 Jun 19. PMID 24953203
- [Derived] Xiao K, Khan F, Link R, Dominguez-Diaz A, Ameyaw P, Alexis J, Tai CH, Assalone V, Nasufi M, Hughes ML, Loeser C, Hung K, Li DK. Efficacy and Safety of Low Volume Bowel Preparation for Colonoscopy in Hospitalized Patients: A Randomized Noninferiority Trial. J Clin Gastroenterol. 2025 Oct 24. doi: 10.1097/MCG.0000000000002269. Online ahead of print. PMID 41128725